CLINICAL TRIAL: NCT02298972
Title: Symptom Support During Chemotherapy: A Mixed Method Study in Adult Patients With Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Flemish League Against Cancer (Other)
Responsible Party: Principal Investigator, Annemarie Coolbrandt, Clinical Nurse Specialist oncology, Universitaire Ziekenhuizen KU Leuven
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B322201422086
Record Dates: First submitted 2014-11-17; First posted 2014-11-24 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Cancer; Chemotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Comparison group (No Intervention): The comparison group will receive standard care.
- Intervention group (Active Comparator): After completion of the comparison group, new patients starting chemotherapy treatment will be offered this study. Study participants will receive the nurse support and selfmanagement intervention.
  Interventions: Behavioral: Nurse support and selfmanagement intervention

INTERVENTIONS:
Behavioral: Nurse support and selfmanagement intervention
  Arms: Intervention group

SUMMARY:
This study evaluates the value of a nursing symptom support en selfmanagement intervention for adult patients with cancer treated with chemotherapy. Using a prospective sequential design with a comparison group who receives standard care and a (later) intervention group who gets the nursing intervention, we will evaluate the effect of this nursing intervention on overall symptom distress (primary outcome) and other measures of symptom burden, self-efficacy, outcome expectations and self-care. By conducting sem-structured interviews with some participants of the intervention group, we will study the patient experience of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients starting first line treatment with (intravenous) chemotherapy
* Ambulatory patients or patients who receive their treatment during short hospital stays
* Regardless of type of cancer, treatment or treatment intention (curative or palliative)
* Who understand sufficiently Dutch to fill out questionnaires
* Who sign informed consent for their participation in the study

Exclusion Criteria:

* Oral anticancer treatment
* Concomitant chemoradiotherapy
* Breast cancer patients who receive nurse counseling throughout their therapy
* Experimental therapy in the context of a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall symptom distress | Longitudinal, during first 3 months after start of treatment
  Summed symptom distress as self-reported on the Symptom Burden Questionnaire
Overall symptom severity | Longitudinal, during first 3 months after start of treatment
  Summed symptom severity as self-reported on the Symptom Burden Questionnaire

SECONDARY OUTCOMES:
Total self-efficacy score | Day 43 of treatment (+/- 1 week)
  Outcome will be measured by a self-report questionnaire: shortened version of the Cancer Behavior Inventory
Total outcome expectations score | Day 43 of treatment (+/- 1 week)
  Outcome will be measured by a self-report questionnaire
Total self-care score | Day 85 of treatment (+/- 1 week)
  Outcome will be measured by a self-report questionnaire: shortened version of the Leuven- Patient Self-care during chemotherapy scale

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium